CLINICAL TRIAL: NCT02223481
Title: A Randomized, Double-blind, Placebo-controlled Evaluation of the Safety and Efficacy of Terbogrel in Patients With Primary Pulmonary Hypertension
Brief Title: Safety and Efficacy of Terbogrel in Patients With Primary Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 528.19
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — terbogrel

ARMS (3):
- Terbogrel low dose (Experimental)
  Interventions: Drug: Terbogrel low dose
- Terbogrel high dose (Experimental)
  Interventions: Drug: Terbogrel high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terbogrel low dose
  Arms: Terbogrel low dose
Drug: Terbogrel high dose
  Arms: Terbogrel high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study sought to determine whether terbogrel was an effective treatment for primary pulmonary hypertension (PPH) by comparing its efficacy and safety to that of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Primary pulmonary hypertension and New York Health Association (NYHA) chronic heart failure (CHF) functional class II-III
* Ability to walk >= 50 meters on the 6 minute walk test
* Resting mean pulmonary artery pressure > 25 mmHg
* Mean right atrial pressure <= 20 mmHg
* Pulmonary capillary wedge pressure <= 15 mmHg
* Cardiac index > 2.5 L/min2
* SvO2 sat. > 63%
* Male of female at least 18 years old
* Signed written informed consent

Exclusion Criteria:

* Secondary pulmonary hypertension due to lung or systemic diseases
* Pregnant of nursing women, or women of childbearing potential who are not using adequate methods of birth control
* Concurrent systematic use of aspirin, aspirin like drugs, or non-steroidal anti-inflammatory drugs (NSAIDs)
* Surgery of bleeding from gastrointestinal, genitourinary tract, cerebrum or retina within past 6 weeks
* History of bleeding diathesis or a platelet count less than 70,000/mm3
* Exercise limited by factors other than fatigue or exertional dyspnea, such as arthritis, claudication, angina, chronic obstructive pulmonary disease, or bronchial asthma
* Myocardial infarction, stroke, or transient ischemic attack within the preceding six months
* Systolic blood pressure < 90 mmHg or > 180 mmHg, or diastolic blood pressure > 110 mmHg
* Known drug or alcohol dependency within one year of entry into the study
* Known hypersensitivity to any component of the study formulation, epoprostenol, nitric oxide, or adenosine
* Psychiatric or other illness or condition which, in the opinion of the principal investigator, may interfere with study participation, compliance, or other elements of the protocol
* Participation in an evaluation of an investigational drug within the past 30 days
* Portal hypertension or cirrhosis of the liver
* Congenital heart disease e.g., atrial septal defect; patent foramen ovale does not exclude patient from the study
* Appetite suppressants such as fenfluramine, dexfenfluramine, and inhibitors of serotonin uptake known to be associated with primary pulmonary hypertension, received within 3 months of entry into the study
* HIV positive
* Vasodilators. Patients will not receive Ca-channel blockers during the study unless the medication was started prior to the study and the patient has been on a stable dose for at least one month prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 1998-05; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Change in distance walked in 6 minutes | baseline, after 3 months of treatment
Change in pulmonary vascular resistance (PVR) | baseline, after 3 months of treatment

SECONDARY OUTCOMES:
Change in pulmonary artery pressure (PAP) | baseline, after 3 months of treatment
Change in cardiac index (CI) | baseline, after 3 months of treatment
Change in venous oxygen saturation (SvO2 sat.) | baseline, after 3 months of treatment
Change in quality of life by SF-36 questionnaire | baseline, after 3 months of treatment
Change in chronic heart failure index | baseline, after 3 months of treatment
  questionnaire
Change in dyspnea/fatigue rating | baseline, after 3 months of treatment